CLINICAL TRIAL: NCT02975947
Title: Effect of Intraoperative Humidified CO2 Insufflation in Open Laparotomy Colorectal Surgery Patients: a Randomized Controlled Trial
Brief Title: Effect of Warmed Humidified CO2 on Peritoneum During Laparotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concord Repatriation General Hospital (Other)
Responsible Party: Principal Investigator, Dr Ju Yong Cheong, Doctor, Concord Repatriation General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HREC/12/CRGH/196
Record Dates: First submitted 2016-11-02; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Peritoneal Inflammation; Peritoneum; Injury
MeSH Terms: conditions — Peritonitis; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Standard intraoperative warming measures including heated blankets, heating with forced warmed air, warming of fluids, and insulation of limbs and head.
  Interventions: Device: Standard heating
- Study Group (Experimental): The study group will receive warmed (37°C), humidified (98% RH) carbon dioxide delivered into the open peritoneal cavity.
  Interventions: Device: Humidified, warmed CO2 insufflation of open peritoneum using Fisher & Paykel's HUMIGARD (Fisher & Paykel Healthcare Ltd, Auckland, New Zealand)

INTERVENTIONS:
Device: Humidified, warmed CO2 insufflation of open peritoneum using Fisher & Paykel's HUMIGARD (Fisher & Paykel Healthcare Ltd, Auckland, New Zealand) — The study group will receive warmed (37°C), humidified (98% RH) carbon dioxide into the open peritoneal cavity using the Fisher & Paykel's HUMIGARD system (Fisher & Paykel Healthcare Ltd, Auckland, New Zealand). This will create a local atmosphere of 100% carbon dioxide (warmed, humidified) in the open peritoneal cavity.
  Arms: Study Group
Device: Standard heating — Standard intraoperative warming measures including heated blankets, heating with forced warmed air, warming of fluids, and insulation of limbs and head
  Arms: Control Group

SUMMARY:
The operating theatre is deliberately made to be cold and dry to prevent bacteria from growing. The problem with this is that during open abdominal surgery, the intestine and the overlying peritoneum is exposed to cold dry air. Surgeons try to stop the bowel/peritoneum from drying by applying warmed saline packs periodically to the bowel. However, this is not always possible. Sometimes, the surgeon has to perform an important component of the procedure (attach bowel/blood vessels together etc) and the bowel/peritoneum visibly dries. When bowel/peritoneum dries damage occurs, inducing inflammation. Inflamed bowel/peritoneum causes the bowel to stick together and form adhesions. Bowel adhesions can cause bowel obstruction. This vicious cycle is repeated when the patient undergoes repetitive open abdominal operations.

This study aimed to be the first human study to:

1. Demonstrate that peritoneal inflammation occurs during open abdominal surgery and also to demonstrate that pro-inflammatory cells (polymorphs, macrophages) are activated during the progress of the operation. This study aims to show that mRNA(using Q-PCR) is increased for pro-inflammatory cytokines. This study also aim to show that proinflammatory cytokines (Interleukin(IL)-1,2,6,9,10, and TNF by ELISA/confirmed using Western Blotting) are elevated during the course of the operation.
2. Demonstrate that the mechanism of bowel/peritoneal inflammation is causally related to the bowel/peritoneum drying (dessication).

This study will attempt to prove this by using humidified, warmed carbon dioxide gas which will warm and moisten the peritoneum/bowel. It is proposed that this will arrest the peritoneal injury and the inflammation. The investigators will attain peritoneal samples during open colorectal operations. The investigators will obtain samples at the beginning and end of the operation. This study design is a randomized controlled trial, where half the patients will receive humidified, warmed carbon dioxide gas during surgery, and the other half will get standard open surgery without carbon dioxide. 40 patients will be recruited in this study. Half (20) will get CO2, and other half (20) will get standard open surgery.

DETAILED DESCRIPTION:
Forty patients undergoing open colorectal surgery will be recruited in this randomized controlled trial.

The study group will receive warmed (37°C), humidified (98% RH) carbon dioxide. The delivered gas will be defined by the United States Pharmacopeia and National Formulary, which requires impurity of less than 200 parts per million, including water vapour. This medical grade CO2 will be warmed to 37°C and humidified to 98% RH using humidification system. The sterility of the system will be assessed regularly as per protocol.

The control group will receive no gas insufflation into the open laparotomy wound. This is current standard practice for all patients undergoing open laparotomy for colorectal resection.

The device that will be used for insufflation of sterile, humidified, warmed CO2 is the Fisher & Paykel's HUMIGARD (Fisher & Paykel Healthcare Ltd, Auckland, New Zealand).

It consists of a bacterial filter and a humidification chamber filed with 180mL sterile water, positioned on a humidifier controller that includes an integrated temperature and flow sensor. The outlet of the humidification chamber is connected to a thermally insulated 2.5m-long heated insufflation tube that maintains temperature and humidity of the gas to its outlet. The warm and humidified CO2 enters a gas diffuser (ST300DF VITA-diffuserTM, Cardia Innovation AB, Stockholm, Sweden) consisting of a 25cm-long polyvinylchloride tube (inner diameter of 2.5mm) with polyurethane foam at its end. The cylindrical polyurethane foam tip diverts the gas jet in multiple directions via the many small paths inside the foam. The gas is thus uniformly distributed and the large diffuser surface area greatly reduces the velocity of the outflow. Thus the system delivers humidified CO2 at 100% relative humidity and 37C to the surgical wound. The gas diffuser will be positioned inside the open abdominal wound cavity (in the right cranial quadrant) at a depth of approximately 4cm from the skin as soon as the abdominal wall retraction has been done. The insufflation of warm humidified CO2 will then start and continue until the abdominal wall retractors are removed and abdominal wall is commenced to be closed.

Calculation of Power: The investigators estimated sample size of 40 patients for 80% power using the literatures' reported standard deviation of levels of 3-chlorotyrosine (which is one of the study's primary biochemical markers of inflammation)

ANALYSIS OF BIOCHEMICAL AND MOLECULAR MARKERS: Where acquired, samples of the human tissue obtained (above) will be homogenised and assigned to biochemistry and molecular analyses. Total RNA will be extracted using a commercial kit, converted to cloned DNA and then probed for various pro-inflammatory genes. Where a change in gene regulation is noted, the investigators will assess the corresponding change in protein level using a combined approach consisting of multiplex ELISA to quantify changes in protein levels and further confirmation with Western blotting using corresponding specific antibodies.

STATISTICAL ANALYSIS: Statistical analysis will be performed using SPSS for Windows version 18.0 GradPack (IBM, New York, USA). Non-parametric continuous variables will be tested using Mann-Whitney U tests and parametric continuous variable will be tested using t-test/ANOVA. Categorical variables will be tested using Fisher exact test.

OUTCOME AND STUDY END POINT:

The study will involve both clinical and laboratory based work, and the outcomes are as follows.

1. Laboratory based work:

   From each patient, 4 samples will be taken and hence 160 samples will be analysed.

   From each sample, the investigators will analyse the activation of pro-inflammatory cells (polymorphs, macrophages), level of messenger RNA.

   The investigators will analyse level of (pro)inflammatory cytokines-- IL1,2,6,9,10, and TNF.

   The investigators will assess the relationship between time (duration of operation) and the inflammatory markers.

   The study will aim to prove that prove that as duration of operation increase, the extent of in inflammation the intestine's surface increases, and that this process can be mitigated by using humidified warmed carbon dioxide gas.
2. Clinical based work:

The study will see whether use of humidified, warmed carbon dioxide gas results in:

* Better core body temperature control
* Less postoperative pain
* Shorter hospital stay
* Less risk of complications, including wound infection, anastomotic leaks.

ELIGIBILITY:
Inclusion Criteria:

* Adults above age 18.
* Elective patients.
* Pathologies: colorectal carcinoma, polyposis syndromes, diverticular diseases, prolapses, and patients with inflammatory bowel disease undergoing elective resection.
* For colorectal carcinoma, all patients whether they are having curative or palliative surgery will be included.
* Patients undergoing open elective colectomy, with or without stoma formation/ bowel anastomosis.

Exclusion Criteria:

* Patients undergoing acute surgery (emergency surgery).
* Patients undergoing Laparoscopic colectomy (multiport, single incision and also hand assisted) as all these patients receive heated humidified CO2.
* For COPD patients, the exclusion criteria would be patients: (1) On home oxygen, (2) Type 2 respiratory failure (CO2 retainers) (3) FEV1<1L, or FEV1/FVC <50% of predicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Inflammatory cytokine level in the peritoneal biopsy samples | At the moment of time when: (1) peritoneal cavity is being opened, (2) when peritoneal cavity is being closed (expected average of 2 hours after peritoneal cavity is first opened)
  Peritoneal samples will be taken when the peritoneal cavity is being opened (at beginning of operation), and also when the peritoneal cavity is being closed (at end of the operation). The change in the level of inflammatory cytokines in between these two time points will be measured
Intraoperative temperature at 30 minutes from start of operation | 30 minutes from start of operation
  Temperature readings during the operation will be taken. Both core body temperature (esophageal) and intraperitoneal temperature will be measured.
Intraoperative temperature at 60 minutes from start of operation | 60 minutes from start of operation
  Temperature readings during the operation will be taken. Both core body temperature (esophageal) and intraperitoneal temperature will be measured.

SECONDARY OUTCOMES:
Postoperative Analgesia requirement for pain | Time from when the patient is moved out of operating theater to when the patient is no longer an inpatient in the hospital ward (discharged), with an expected average of 1 week
  Postoperative pain as measured by MEDD (Morphine Equivalent Daily Dose)
Length of in-patient hospital stay | duration of hospital stay, an expected average of 1 week
  number of days patient stayed postoperatively in hospital
Anastomotic leaks | 6 months
  The occurrence of anastomotic leak in the 6 months after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Concord Repatriation General Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Persson M, van der Linden J. Intraoperative CO2 insufflation can decrease the risk of surgical site infection. Med Hypotheses. 2008;71(1):8-13. doi: 10.1016/j.mehy.2007.12.016. Epub 2008 Mar 4. PMID 18304752
- [Result] Persson M, van der Linden J. Can wound desiccation be averted during cardiac surgery? An experimental study. Anesth Analg. 2005 Feb;100(2):315-320. doi: 10.1213/01.ANE.0000140243.97570.DE. PMID 15673849
- [Result] Persson M, Elmqvist H, van der Linden J. Topical humidified carbon dioxide to keep the open surgical wound warm: the greenhouse effect revisited. Anesthesiology. 2004 Oct;101(4):945-9. doi: 10.1097/00000542-200410000-00020. PMID 15448528
- [Result] Persson M, Svenarud P, Flock JI, van der Linden J. Carbon dioxide inhibits the growth rate of Staphylococcus aureus at body temperature. Surg Endosc. 2005 Jan;19(1):91-4. doi: 10.1007/s00464-003-9334-z. Epub 2004 Nov 11. PMID 15529188
- [Result] Persson M, van der Linden J. Wound ventilation with ultraclean air for prevention of direct airborne contamination during surgery. Infect Control Hosp Epidemiol. 2004 Apr;25(4):297-301. doi: 10.1086/502395. PMID 15108726
- [Result] Svenarud P, Persson M, Van Der Linden J. Efficiency of a gas diffuser and influence of suction in carbon dioxide deairing of a cardiothoracic wound cavity model. J Thorac Cardiovasc Surg. 2003 May;125(5):1043-9. doi: 10.1067/mtc.2003.50. PMID 12771877
- [Result] Svenarud P, Persson M, van der Linden J. Intermittent or continuous carbon dioxide insufflation for de-airing of the cardiothoracic wound cavity? An experimental study with a new gas-diffuser. Anesth Analg. 2003 Feb;96(2):321-7, table of contents. doi: 10.1097/00000539-200302000-00005. PMID 12538172
- [Result] Hannenberg AA, Sessler DI. Improving perioperative temperature management. Anesth Analg. 2008 Nov;107(5):1454-7. doi: 10.1213/ane.0b013e318181f6f2. No abstract available. PMID 18931198
- [Result] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Result] Insler SR, Sessler DI. Perioperative thermoregulation and temperature monitoring. Anesthesiol Clin. 2006 Dec;24(4):823-37. doi: 10.1016/j.atc.2006.09.001. PMID 17342966
- [Result] Sessler DI. Non-pharmacologic prevention of surgical wound infection. Anesthesiol Clin. 2006 Jun;24(2):279-97. doi: 10.1016/j.atc.2006.01.005. PMID 16927930
- [Result] Binda MM, Koninckx PR. Prevention of adhesion formation in a laparoscopic mouse model should combine local treatment with peritoneal cavity conditioning. Hum Reprod. 2009 Jun;24(6):1473-9. doi: 10.1093/humrep/dep053. Epub 2009 Mar 3. PMID 19258346
- [Result] Tsuchiya M, Sato EF, Inoue M, Asada A. Open abdominal surgery increases intraoperative oxidative stress: can it be prevented? Anesth Analg. 2008 Dec;107(6):1946-52. doi: 10.1213/ane.0b013e318187c96b. PMID 19020142
- [Result] Peng Y, Zheng M, Ye Q, Chen X, Yu B, Liu B. Heated and humidified CO2 prevents hypothermia, peritoneal injury, and intra-abdominal adhesions during prolonged laparoscopic insufflations. J Surg Res. 2009 Jan;151(1):40-7. doi: 10.1016/j.jss.2008.03.039. Epub 2008 Apr 23. PMID 18639246
- [Result] Brokelman WJ, Holmdahl L, Bergstrom M, Falk P, Klinkenbijl JH, Reijnen MM. Heating of carbon dioxide during insufflation alters the peritoneal fibrinolytic response to laparoscopic surgery : A clinical trial. Surg Endosc. 2008 May;22(5):1232-6. doi: 10.1007/s00464-007-9597-x. Epub 2007 Oct 18. PMID 17943363
- [Result] Ivarsson ML, Bergstrom M, Eriksson E, Risberg B, Holmdahl L. Tissue markers as predictors of postoperative adhesions. Br J Surg. 1998 Nov;85(11):1549-54. doi: 10.1046/j.1365-2168.1998.00859.x. PMID 9823923
- [Result] Moehrlen U, Ziegler U, Boneberg E, Reichmann E, Gitzelmann CA, Meuli M, Hamacher J. Impact of carbon dioxide versus air pneumoperitoneum on peritoneal cell migration and cell fate. Surg Endosc. 2006 Oct;20(10):1607-13. doi: 10.1007/s00464-005-0775-4. Epub 2006 Jul 3. PMID 16823647
- [Result] Erikoglu M, Yol S, Avunduk MC, Erdemli E, Can A. Electron-microscopic alterations of the peritoneum after both cold and heated carbon dioxide pneumoperitoneum. J Surg Res. 2005 May 1;125(1):73-7. doi: 10.1016/j.jss.2004.11.029. PMID 15836853
- [Result] Enfors SO, Molin G. The influence of high concentrations of carbon dioxide on the germination of bacterial spores. J Appl Bacteriol. 1978 Oct;45(2):279-85. doi: 10.1111/j.1365-2672.1978.tb04223.x. No abstract available. PMID 31348
- [Result] Ott DE. Correction of laparoscopic insufflation hypothermia. J Laparoendosc Surg. 1991 Aug;1(4):183-6. doi: 10.1089/lps.1991.1.183. PMID 1834266
- [Result] Frank SM, Beattie C, Christopherson R, Norris EJ, Perler BA, Williams GM, Gottlieb SO. Unintentional hypothermia is associated with postoperative myocardial ischemia. The Perioperative Ischemia Randomized Anesthesia Trial Study Group. Anesthesiology. 1993 Mar;78(3):468-76. doi: 10.1097/00000542-199303000-00010. PMID 8457047
- [Result] Schmied H, Kurz A, Sessler DI, Kozek S, Reiter A. Mild hypothermia increases blood loss and transfusion requirements during total hip arthroplasty. Lancet. 1996 Feb 3;347(8997):289-92. doi: 10.1016/s0140-6736(96)90466-3. PMID 8569362
- [Result] Hazebroek EJ, Schreve MA, Visser P, De Bruin RW, Marquet RL, Bonjer HJ. Impact of temperature and humidity of carbon dioxide pneumoperitoneum on body temperature and peritoneal morphology. J Laparoendosc Adv Surg Tech A. 2002 Oct;12(5):355-64. doi: 10.1089/109264202320884108. PMID 12470410
- [Derived] Cheong JY, Chami B, Fong GM, Wang XS, Keshava A, Young CJ, Witting P. Randomized clinical trial of the effect of intraoperative humidified carbon dioxide insufflation in open laparotomy for colorectal resection. BJS Open. 2020 Feb;4(1):45-58. doi: 10.1002/bjs5.50227. Epub 2019 Nov 17. PMID 32011809